CLINICAL TRIAL: NCT05209776
Title: Local Inflammation in Arrhythmogenic Right Ventricular Cardiomyopathy
Acronym: LI-ARVC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/21/0026
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Arrhythmogenic Right Ventricular Dysplasia
Keywords: Cardiac Electrophysiologic Techniques; Inflammation; Cytokines; Interleukin-1; Interleukin-6; Interleukin-10; Transforming Growth Factor beta; Tumor Necrosis Factor-alpha
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Inflammation; Camurati-Engelmann Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Carrier of a definite diagnosis of arrhythmogenic dysplasia of the right ventricle in line with the criteria of the Task Force 2010 (see Appendices), admitted for an electrical mapping of the right ventricle
  Interventions: Biological: Peripheral immunological assessment on venous blood; Biological: Immunological assessment carried out on intracardiac material
- Control case (Experimental): Without heart disease, admitted for a Kent bundle ablation or endocavity procedure / Wolff-Parkinson-White syndrome or common flutter (in subjects in whom the same irrigated material will be used and for whom echocardiography will have excluded associated heart disease).
  Interventions: Biological: Peripheral immunological assessment on venous blood; Biological: Immunological assessment carried out on intracardiac material

INTERVENTIONS:
Biological: Peripheral immunological assessment on venous blood — Peripheral immunological assessment carried out as part of the research, on venous blood at the puncture point necessary for the electrophysiological examination: 1 heparin tube and 1 EDTA tube
Biological: Immunological assessment carried out on intracardiac material — Immunological assessment carried out as part of the research, on intracardiac material taken during the electrophysiological examination: 1 EDTA tube

SUMMARY:
The understanding of ARVC pathophysiology remains incomplete. Several clues indicate that disease progression is mediated through inflammation. The present study aim to document the feasibility of detecting the potential presence of intracardiac local inflammatory components in patients with ARVC.

DETAILED DESCRIPTION:
Arrhythmogenic right ventricular cardiomyopathy (ARVC) is a heritable condition characterized by right ventricular (RV) dilatation/dysfunction and malignant ventricular arrhythmias. The understanding of ARVC pathophysiology remains incomplete. Several clues indicate that disease progression is mediated through inflammation. First, presence of subepicardial late gadolinium enhancement sharing the same characteristics as the ones found in myocarditis is common on cardiac magnetic resonance imaging (CMR). Second, clinical pathology findings of inflammatory infiltrates of mononuclear cells are frequent and correlate to the extent and severity of ARVC. Finally, from a biological standpoint, the exploratory study conducted by Campian et al. has shown an exaggerated humoral inflammatory response in peripheral blood whilst anti-desmoglein-2 antibodies (targeting a component of the desmosome) emerge as a sensitive and specific biomarker for ARVC. As specific treatments for ARVC are currently lacking, a better understanding of the humoral pathophysiology of the disease could unlock new therapeutic targets. We recently demonstrated that collecting local cardiomyocytes was feasible through irrigated ablation catheters in patients with ARVC. These steerable catheters may easily map the whole right ventricle and locate endocardial or epicardial scars. Aspiration of local blood or cellular material through the inner lumen of the catheter once pressed on the parietal wall may be an interesting technique for retrieving local inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* For cases:

  * Arrhythmogenic right ventricular dysplasia diagnosed (according to 2010 Task Force Criteria)
  * Admitted for right ventricle electrophysiologic mapping
* For controls * Admitted for ablation procedures (accessory pathway, atrial flutter) on otherwise healthy hearts.

Exclusion Criteria:

* Diagnostic of systemic chronic inflammatory disease
* Presence of possible or proven cardiac involvement of an inflammatory disease, an acute or chronic infectious disease.
* Taking immunosuppressant or immunomodulating medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Identify the inflammatory components by C-reactive protein | 24 months
  Rate of C-reactive protein in the blood
Identify the inflammatory components by interleukine1 | 24 months
  Rate of interleukin 1 beta in the blood
Identify the inflammatory components by onterleukine6 | 24 months
  Rate of interleukin 6 in the blood
Identify the inflammatory components by interleukine10 | 24 months
  Rate of interleukin 10 in the blood
Identify the inflammatory components by Tumor Necrosis Factor | 24 months
  Rate of Tumor Necrosis Factor alpha in the blood
Identify the inflammatory components by Transforming Growth Factor | 24 months
  Rate of Transforming Growth Factor beta in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAURY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital Center, Toulouse, France

IPD SHARING:
Plan to Share IPD: No